CLINICAL TRIAL: NCT05227625
Title: Randomized Controlled Trial Assessing the Effectiveness of a Psychological Management Program for Body Dissatisfaction in Eating Disorders
Brief Title: Randomized Study Assessing a Program of Body Dissatisfaction Psychological Care in Eating Disorders
Acronym: INCCA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RECHMPL21_0279
Record Dates: First submitted 2022-01-26; First posted 2022-02-07 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Eating Disorders
Keywords: eating disorders; anorexia; bulimia; body dissatisfaction
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia; Bulimia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Body dissatisfaction management group (Experimental): ACT-inspired group for the management of body dissatisfaction
  Interventions: Behavioral: body dissatisfaction management group
- relaxation group (Active Comparator): standardized relaxation program
  Interventions: Behavioral: Relaxation Group

INTERVENTIONS:
Behavioral: body dissatisfaction management group — Our group is composed of 10 weekly session of 2 hours led by a psychologist trained in the management of ED and ACT therapy.
  Each group will be composed of 5 to 10 people. First of all, the group will lead the participants to better know and understand the impact of BD on the symptomatology of ED by teaching current scientific knowledge on the subject. In a second step, the group will guide the patients in the acquisition of psychological skills to deal with events related to BD and to engage in actions towards the values that give meaning to their existence.
  Arms: Body dissatisfaction management group
Behavioral: Relaxation Group — Participants will be included in a standardized relaxation program consisting of a weekly 2 hour session for 10 weeks. The group will be led by a psychologist trained in relaxation and in particular in abdominal and muscular relaxation techniques. Each group will be composed of 5 to 10 people. Initially, the therapy will lead the participants to recognize the signs of anxiety and to understand the physiological mechanisms involved. Classic techniques of anxiety management will then be introduced (cardiac coherence, abdominal and muscular relaxation, Jacobson technique, Schultz autogenic training). These techniques will be tested in session. Participants will be encouraged to practice these techniques at home.
  Arms: relaxation group

SUMMARY:
Eating disorders (ED) are a major public health problem for which current treatments are insufficiently effective. The transdiagnostic approach of eating disorders highlights body dissatisfaction (BD) as a major factor in the development and maintenance of the different types of eating disorders. Thus, we hypothesize that a group focused on the management of BDc would improve the prognosis of patients with eating disorders.

DETAILED DESCRIPTION:
Main and secondary objectives: To evaluate the effectiveness of a BD management group on the level of body dissatisfaction in patients suffering from an ED (BSQ-34 total score immediately after intervention). Secondary: To assess the effectiveness of a BD management group in 1) reducing the desire for thinness, 2) improving quality of life, 3) improving ED symptoms, 4) improvement in depressive symptomatology, 5) increase in cognitive flexibility and acceptance of unpleasant psychological events, 6) improvement in overall functioning.

Methodology : Open randomized controlled trial with two intervention arms (management of BD versus relaxation). Main inclusion criteria: patients over 16 years of age suffering from an ED, presenting moderate to severe BD (BSQ-34≥111) and normal BMI

Main endpoint: evolution of the level of BD (BSQ-34) immediately after the intervention. Secondary judgment criteria: change in the level of BD (BSQ-34) at 1 and 3 months post-intervention & change in eating symptomatology (EDI, EDE-Q), quality of life (EDQOL), level of depression (MADRS), cognitive flexibility ( AAQ), functioning (WSAS) immediately post-intervention, at 1 and 3 months post-intervention.

Procedure: The participation of each patient includes 4 evaluation visits: inclusion, just after the end of the intervention, at 1 and 3 months after the end of the intervention

Benefits / prospects: We hope that patients who have integrated the interventional group will show a significant improvement in their BD, their functioning and the overall prognosis of the disorder. Positive results would permit to consider a larger multicenter study evaluating the long-term effect of the group on different dimensions of the ED. Finally, it would then be possible to offer standardized care that can be generalized to other centers.

ELIGIBILITY:
Inclusion Criteria:

* ED according to DSM 5 criteria (all types of ED can be included: anorexia, bulimia, binge eating disorder, atypical ED, etc.)
* BMI between 18.5 kg/m2 and 24.9 kg/m2).
* woman over the age of 16
* moderate to severe body dissatisfaction (total BSQ score greater than or equal to 111)

Exclusion Criteria:

* current severe psychiatric pathology other than the TCA (severe depression, schizophrenia, etc.) which may alter the ability to follow the group in the opinion of the investigator
* Patient under legal protection measure (guardianship, curatorship, safeguard of justice, authorization family or future protection mandate activated
* Pregnant or breastfeeding women according
* Patient not affiliated to a social security scheme, or beneficiary of such a scheme
* Patient unable to understand the nature, purpose and methodology of the study
* Patient who did not sign the informed consent
* Patient whose legal guardian has not given consent to inclusion

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Body dissatisfaction | immediate post intervention
  Assessment of body dissatisfaction using Body shape questionnaire (BSQ-34) 34-item self-administered questionnaire assessing body dissatisfaction across four dimensions: avoidance and social shame of body exposure, body dissatisfaction with lower parts of the body, use of laxatives and vomiting to reduce body dissatisfaction, cognitions and maladaptive behaviors to control weight. The total score ranges from 0 to 204. A score below 80 indicates no excessive body dissatisfaction, a score between 80 and 100 indicates mild body dissatisfaction, between 111 and 140 moderate body dissatisfaction and a score above 140 indicates severe body dissatisfaction

SECONDARY OUTCOMES:
Body dissatisfaction | 1 month post intervention
  Assessment of body dissatisfaction using Body shape questionnaire (BSQ-34) 34-item self-administered questionnaire assessing body dissatisfaction across four dimensions: avoidance and social shame of body exposure, body dissatisfaction with lower parts of the body, use of laxatives and vomiting to reduce body dissatisfaction, cognitions and maladaptive behaviors to control weight. The total score ranges from 0 to 204. A score below 80 indicates no excessive body dissatisfaction, a score between 80 and 100 indicates mild body dissatisfaction, between 111 and 140 moderate body dissatisfaction and a score above 140 indicates severe body dissatisfaction
Body dissatisfaction | 3 months post intervention
  Assessment of body dissatisfaction using Body shape questionnaire (BSQ-34) 34-item self-administered questionnaire assessing body dissatisfaction across four dimensions: avoidance and social shame of body exposure, body dissatisfaction with lower parts of the body, use of laxatives and vomiting to reduce body dissatisfaction, cognitions and maladaptive behaviors to control weight. The total score ranges from 0 to 204. A score below 80 indicates no excessive body dissatisfaction, a score between 80 and 100 indicates mild body dissatisfaction, between 111 and 140 moderate body dissatisfaction and a score above 140 indicates severe body dissatisfaction
eating behavior | immediate post intervention
  Assessment of eating behavior using Eating disorder Inventory (EDI-2). 91-item self-questionnaire aim to evaluate food-related attitudes and behaviors. 11 dimensions emerge : search for thinness, bulimia, dissatisfaction with the body, inefficiency, perfectionism, interpersonal mistrust, interoceptive awareness, fear of maturity, asceticism, impulse control, social insecurity.
  A high score reflects a higher intensity of symptoms
eating behavior | 1 month post intervention
  Assessment of eating behavior using Eating disorder Inventory (EDI-2). 91-item self-questionnaire aim to evaluate food-related attitudes and behaviors. 11 dimensions emerge : search for thinness, bulimia, dissatisfaction with the body, inefficiency, perfectionism, interpersonal mistrust, interoceptive awareness, fear of maturity, asceticism, impulse control, social insecurity.
  A high score reflects a higher intensity of symptoms
eating behavior | 3 months post intervention
  Assessment of eating behavior using Eating disorder Inventory (EDI-2) 91-item self-questionnaire aim to evaluate food-related attitudes and behaviors. 11 dimensions emerge : search for thinness, bulimia, dissatisfaction with the body, inefficiency, perfectionism, interpersonal mistrust, interoceptive awareness, fear of maturity, asceticism, impulse control, social insecurity.
  A high score reflects a higher intensity of symptoms
Quality of life level | immediate post intervention
  Assessment of quality of life using the Eating Disorder Quality Of Life (EDQOL).
  EDQOL is a self-questionnaire assessing the quality of life, specific to eating disorders. 4 dimensions are assessed: Psychological, Physical/Cognitive, Financial, Work/School. The scale also produces an overall score. The higher the score, the more the eating disorder impacts the patient's quality of life
Quality of life level | 1 month post intervention
  Assessment of quality of life using the Eating Disorder Quality Of Life (EDQOL).
  EDQOL is a self-questionnaire assessing the quality of life, specific to eating disorders. 4 dimensions are assessed: Psychological, Physical/Cognitive, Financial, Work/School. The scale also produces an overall score. The higher the score, the more the eating disorder impacts the patient's quality of life
Quality of life level | 3 months post intervention
  Assessment of quality of life using the Eating Disorder Quality Of Life (EDQOL).
  EDQOL is a self-questionnaire assessing the quality of life, specific to eating disorders. 4 dimensions are assessed: Psychological, Physical/Cognitive, Financial, Work/School. The scale also produces an overall score. The higher the score, the more the eating disorder impacts the patient's quality of life
Eating disorder symptomatology | immediate post intervention
  Assessment of Eating disorder symptomatology using the Eating disorder Examination (EDE-q). Self-administered questionnaire assessing the intensity of eating symptoms over the past 28 days. A total score as well as 4 sub-scores (restriction, diet, weight, shape) varying from 0 to 6. The higher the score, the more severe the symptoms.
Eating disorder symptomatology | 1 month post intervention
  Assessment of Eating disorder symptomatology using the Eating disorder Examination (EDE-q). Self-administered questionnaire assessing the intensity of eating symptoms over the past 28 days. A total score as well as 4 sub-scores (restriction, diet, weight, shape) varying from 0 to 6. The higher the score, the more severe the symptoms.
Eating disorder symptomatology | 3 months post intervention
  Assessment of Eating disorder symptomatology using the Eating disorder Examination (EDE-q). Self-administered questionnaire assessing the intensity of eating symptoms over the past 28 days. A total score as well as 4 sub-scores (restriction, diet, weight, shape) varying from 0 to 6. The higher the score, the more severe the symptoms.
depressive symptomatology | immediate post intervention
  Assessment of depressive symptomatology using Montgomery Asberg Depression Scale (MADRS). This hetero-questionnaire assesses the intensity of the patient's depressive symptoms. The total score between 0 and 60 corresponds to the sum of the 10 items. The higher the score, the more severe the symptoms.
depressive symptomatology | 1 month post intervention
  Assessment of depressive symptomatology using Montgomery Asberg Depression Scale (MADRS). This hetero-questionnaire assesses the intensity of the patient's depressive symptoms. The total score between 0 and 60 corresponds to the sum of the 10 items. The higher the score, the more severe the symptoms.
depressive symptomatology | 3 months post intervention
  Assessment of depressive symptomatology using Montgomery Asberg Depression Scale (MADRS). This hetero-questionnaire assesses the intensity of the patient's depressive symptoms. The total score between 0 and 60 corresponds to the sum of the 10 items. The higher the score, the more severe the symptoms.
cognitive flexibility | immediate post intervention
  Assessment of cognitive flexibility using the Acceptance and Action Questionnaire (AAQ).
  the AAQ is 7-item self-questionnaire to assess psychological flexibility and psychological acceptance
cognitive flexibility | 1 month post intervention
  Assessment of cognitive flexibility using the Acceptance and Action Questionnaire (AAQ).
  the AAQ is 7-item self-questionnaire to assess psychological flexibility and psychological acceptance
cognitive flexibility | 3 months post intervention
  Assessment of cognitive flexibility using the Acceptance and Action Questionnaire (AAQ).
  the AAQ is 7-item self-questionnaire to assess psychological flexibility and psychological acceptance
Global functioning | immediate post intervention
  Assessment of Global functioning using the Work and Social Adjustment Scale . The WSAS is self-questionnaire of 5 items aimed at evaluating the consequences of the ED on the overall functioning of the patient. Each item is rated from 0 to 8. The score of the scale therefore varies from 0 (no functioning problem) to 40 (maximum problems). A score greater than 20 suggests a significant impairment in functioning. A score between 10 and 20 suggests moderate impairment. A score of less than 10 suggests no functioning problem
Global functioning | 1 month post intervention
  Assessment of Global functioning using the Work and Social Adjustment Scale . The WSAS is self-questionnaire of 5 items aimed at evaluating the consequences of the ED on the overall functioning of the patient. Each item is rated from 0 to 8. The score of the scale therefore varies from 0 (no functioning problem) to 40 (maximum problems). A score greater than 20 suggests a significant impairment in functioning. A score between 10 and 20 suggests moderate impairment. A score of less than 10 suggests no functioning problem
Global functioning | 3 months post intervention
  Assessment of Global functioning using the Work and Social Adjustment Scale . The WSAS is self-questionnaire of 5 items aimed at evaluating the consequences of the ED on the overall functioning of the patient. Each item is rated from 0 to 8. The score of the scale therefore varies from 0 (no functioning problem) to 40 (maximum problems). A score greater than 20 suggests a significant impairment in functioning. A score between 10 and 20 suggests moderate impairment. A score of less than 10 suggests no functioning problem
mindfulness skills | immediate post intervention
  Assessment of mindfulness skills using Mindful Attention Awarness Scale (MAAS). 15-item self-questionnaire to assess spontaneous mindfulness skills.
mindfulness skills | 1 month post intervention
  Assessment of mindfulness skills using Mindful Attention Awarness Scale (MAAS). 15-item self-questionnaire to assess spontaneous mindfulness skills.
mindfulness skills | 3 months post intervention
  Assessment of mindfulness skills using Mindful Attention Awarness Scale (MAAS). 15-item self-questionnaire to assess spontaneous mindfulness skills.